CLINICAL TRIAL: NCT06888271
Title: DNA Methylation in Brugada Syndrome and Risk of Sudden Cardiac Death (ANDROMEDA)
Brief Title: DNA Methylation in Brugada Syndrome and Risk of Sudden Cardiac Death
Acronym: ANDROMEDA
Status: Not yet recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Responsible Party: Principal Investigator, Giuditta Benincasa, Principal Investigator, University of Campania Luigi Vanvitelli
Other Study IDs: Vanvitelli-Benincasa G; PE00000015 (Other Grant/Funding Number: National Recovery and Resilience Plan (NRRP))
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Brugada Syndrome; Sudden Cardiac Death Due to Cardiac Arrhythmia
Keywords: DNA methylation; Liquid biopsy; Sudden cardiac death; Brugada syndrome
MeSH Terms: conditions — Brugada Syndrome; Death, Sudden, Cardiac

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Healthy subjects: The control group consisted of unrelated age- and sex-matched healthy subjects as volunteer blood donors with no evidence of any ECG abnormalities, inherited arrhythmia, genetic cardiomyopathy, and no history of ventricular arrhythmia, unexplained syncope, unexplained sudden cardiac arrest/ death.
- Brugada patients: Brugada syndrome was confirmed when the 12-lead ECG showed ST-segment elevation with a type-1 morphology of ≥2 mm in ≥1 right precordial lead either spontaneously or after a provocative drug test (intravenous administration of a Class I antiarrhythmic) in the absence of any structural heart disease.

SUMMARY:
The goal of this observational study is to evaluate if there are differences in DNA methylation of peripheral blood in patients with Brugada syndrome and healthy subjects. The main question it aims to answer is:

Does DNA methylation changes distinguish Brugada patients from healthy controls?

Does DNA methylation changes distinguish Brugada patients with high versus low risk of sudden cardiac death?

DETAILED DESCRIPTION:
The Investigators will enroll 10 patients with Brugada syndrome and 10 age and sex matched healthy controls. We will collect 5 mL of peripheral blood and will analyze genome-wide DNA methylation via EPIC array platform. Bioinformatic algorithms and network analysis will be applied to identify possible diagnostic and predictive biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Brugada syndrome was confirmed when the 12-lead ECG showed ST-segment elevation with a type-1 morphology of ≥2 mm in ≥1 right precordial lead either spontaneously or after a provocative drug test (intravenous administration of a Class I antiarrhythmic) in the absence of any structural heart disease.
* >18 years
* Unrelated patients

Exclusion Criteria:

* Related patients
* Not type 1 Br patter

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with Brugada syndrome attended the Cardiology Dept. at University of Campania "L. Vanvitelli", Monaldi Hospital (Naples, Italy). The control group consisted of unrelated age- and sex-matched healthy subjects as volunteer blood donors attending the U.O.C. Divisione di Immunologia Clinica, Immunoematologia, Medicina Trasfusionale at University of Campania "L. Vanvitelli" (Naples, Italy).
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of differentially methylated genes as assessed by EPIC microarray | 3 months
  We will compare the methylation profiles of patients and controls in order to obtain a panel of differentially methylated genes.

SECONDARY OUTCOMES:
Diagnostic performance of differentially methylated regions predicting the risk of sudden cardiac death | 6 months
  We will perform a subgroup analysis of Brugada patients (high vs. low risk of sudden cardiac death). ROC curve analysis will be performed to identify which differentially methylated genese may be useful to predict the risk of sudden cardiac death.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Benincasa G, Pepin ME, Russo V, Cacciatore F, D'Alto M, Argiento P, Romeo E, Chiappetti R, Laezza N, Wende AR, Schiattarella GG, Coscioni E, La Montagna A, Amarelli C, Maiello C, Golino P, Condorelli G, Napoli C. High-resolution DNA methylation changes reveal biomarkers of heart failure with preserved ejection fraction versus reduced ejection fraction. Basic Res Cardiol. 2025 Apr;120(2):347-361. doi: 10.1007/s00395-024-01093-7. Epub 2024 Dec 27. PMID 39725721